CLINICAL TRIAL: NCT00361088
Title: A Dose Escalation of Zarnestra (R115777) Combined With Velcade® (PS-341) in Patients With Relapsed Multiple Myeloma
Brief Title: A Combination of Zarnestra With Velcade for Patients With Relapsed Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Initial Principal Investigator left Moffitt
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Melissa Alsina, H. Lee Moffitt Cancer Center and Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13971; 7032 (Other: NCI)
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2011-05

CONDITIONS: Multiple Myeloma
Keywords: Velcade (PS-341); Bortezomib; Zarnestra (R115777); Tipifarnib
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I (Experimental)
  Interventions: Drug: PS-341; Drug: R11577
- Phase II (Experimental)
  Interventions: Drug: PS-341; Drug: R11577

INTERVENTIONS:
Drug: PS-341 — Phase I and II: 1.3mg/m2 iv days 1,4,8,11
  Other Names: bortezomib; Velcade®
Drug: R11577 — Phase I: 100mg po BID days 1014 for Cohort 1, 200mg po BID days 1014 for Cohort 2, 300mg po BID days 1014 for Cohort 3.
  Phase II: Maximum Tolerated Dose (MTD)
  Other Names: Zarnestra

SUMMARY:
In Phase I, patients will receive a combination of PS-341 (Velcade) and R115777 (Zarnestra) to determine the dose limiting toxicity (DLT). Once DLT is determined, patients in Phase II will be receive the maximum tolerated dose (MTD) to complete 8 cycles of therapy. Treatment will continue if there is evidence of continued response for 8 cycles. Patients will receive follow up to include normal laboratory evaluations at least every 3 months and a skeletal survey will be performed at least every 6 months.

DETAILED DESCRIPTION:
In Phase I, patients will receive intravenous PS-341 (Velcade) and 3 different dose levels of oral R115777 (Zarnestra). Dose Limiting Toxicity (DLT) will be determined over a period of one cycle and dose escalation to the next level will not occur until all patients projected at each level complete one cycle of therapy. Once DLT is determined, patients in Phase I and all patients enrolled for the phase II component will be treated at the maximum tolerated dose (MTD) to complete 8 cycles of therapy. Treatment will continue beyond 8 cycles if there is evidence of continued response. The study regimen will consist of two weeks of treatment followed by one week off for a total cycle duration of three weeks. If disease stabilization occurs (noted on 2 consecutive cycles) after the standard 8 cycles are given, treatment will be discontinued.

Patients are to be monitored for adverse events throughout the treatment phases and for a minimum of 30 days after their last dose of drugs. Follow up will include history and physical exam with laboratory evaluation at least every 3 months. Laboratories will include CMP, CBC, SPEP, UPEP, and quantitative immunoglobulins. A skeletal survey will be performed at least every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent
* Female subject is either post-menopausal/surgically sterilized or willing to use an acceptable method of birth control for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* Diagnosis of stage II or III multiple myeloma and have relapsed after at least one prior therapies confirmed by the presence of:

  1. A new lytic lesion
  2. A 25% increase in urine or serum monoclonal protein
* Patient can have received PS-341 (Velcade) previously and does not require a previous response.
* Patients must have measurable disease. One or more of the following must be present to qualify for this study:

  1. Serum M-component greater than or equal to 1.0 gm/dl (10.0 g/L) by serum protein electrophoresis
  2. Urine M-protein excretion > 200 mg/24 (0.2 g/24h) hours, by urine protein electrophoresis
  3. Abnormal serum free light chain ratio with elevated Kappa or Lambda light chains in serum
* Baseline measurements must be done within 21 days of study entry.
* Karnofsky Performance Status Scale > 60.
* Greater than or equal to 18 years of age.
* Expected survival of greater than 8 weeks.
* Swallow intact study medication tablets.
* Can follow directions or has a caregiver who will be responsible for administering study medication.

Exclusion Criteria:

* Previously treated with R115777 (Zarnestra).
* Undergone an allogeneic bone marrow transplant.
* A platelet count of <100,000 x 10 to the 9 power/L within 14 days before enrollment.
* Absolute neutrophil count of <1.0 x 10 to the 9 power/L within 14 days before enrollment.
* Measured creatinine > 1.5 X the upper limits of normal within 14 days before enrollment.
* Greater than or equal to Grade 2 peripheral neuropathy within 14 days before enrollment.
* Hypersensitivity to bortezomib, boron, mannitol or imidazole compounds
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening.
* Received other investigational drugs within 14 days of enrollment or immunotherapy within 30 days of enrollment.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Ongoing radiation therapy or radiation therapy within 14 days prior to first treatment.
* Cytotoxic chemotherapy within 30 days prior to first treatment.
* Therapy with high-dose corticosteroids within 14 days prior to first treatment.
* Presence of any of the following excludes a patient from entering the study until such condition is resolved (determined within 14 days prior to the first treatment):

  1. Elevated total bilirubin > 2mg/dl, or direct bilirubin > 2 times the ULN.
  2. Serum glutamic oxaloacetic transaminase (AST, formerly SGOT) or serum glutamic pyruvic transaminase (ALT, formerly SGPT) > 2 times the ULN
  3. Serum calcium > 12 mg/dL.
  4. Concurrent serious infection.
  5. Life-threatening illness (unrelated to tumor).
* History of any other ACTIVE and INVASIVE cancer other than the present condition (except non-melanoma skin cancer), unless in complete remission and off of all therapy for that disease for a minimum of 3 years.
* Prohibited/allowable medications or precautions:

  1. Enzyme-inducing anti-epileptic medications (e.g. phenytoin, phenobarbital, carbamazepine) are not allowed.
  2. Non-enzyme anti-epileptic medications will be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Average of 6 months
  Determine the dose limiting toxicity at 3 weeks post treatment
Maximum Tolerated Dose | Average of 6 months
  Determine the maximum tolerated dose
Response Rates | Average of 6 months
  Determine response rates after 8 cycles of treatment
Toxicity | Average of 6 months
  Determine toxicity profiles

SECONDARY OUTCOMES:
Progression Free Survival | Average of 12 months
  Determine progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Alsina, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States